CLINICAL TRIAL: NCT01668927
Title: Helicobacter Pylori Treatment
Brief Title: Empirical Rescue Therapies of Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Dr. HONG LU, professor of GI Division, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjkls_2012009
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Functional Dyspepsia; Scarred Peptic Ulcer
MeSH Terms: interventions — Proton Pump Inhibitors; Lansoprazole; Bismuth; Metronidazole; Tetracycline; Furazolidone; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- tetracycline/furazolidone (Experimental): one of the four empirical rescue therapies
  Interventions: Drug: Proton Pump Inhibitor; Drug: Bismuth; Drug: Tetracycline; Drug: Furazolidone
- amoxicillin/tetracycline (Experimental): one of the four empirical rescue therapies
  Interventions: Drug: Proton Pump Inhibitor; Drug: Bismuth; Drug: Tetracycline; Drug: Amoxicillin
- amoxicillin/furazolidone (Experimental): one of the four empirical rescue therapies
  Interventions: Drug: Proton Pump Inhibitor; Drug: Bismuth; Drug: Furazolidone; Drug: Amoxicillin
- tetracycline /metronidazole (Active Comparator): Classical rescue therapy
  Interventions: Drug: Proton Pump Inhibitor; Drug: Bismuth; Drug: Metronidazole; Drug: Tetracycline

INTERVENTIONS:
Drug: Proton Pump Inhibitor
  Other Names: Lansoprazole
Drug: Bismuth
  Other Names: Bismuth potassium citrate
Drug: Metronidazole
  Arms: tetracycline /metronidazole
Drug: Tetracycline
  Arms: amoxicillin/tetracycline; tetracycline /metronidazole; tetracycline/furazolidone
Drug: Furazolidone
  Arms: amoxicillin/furazolidone; tetracycline/furazolidone
Drug: Amoxicillin
  Arms: amoxicillin/furazolidone; amoxicillin/tetracycline

SUMMARY:
The increase of antibiotic resistance to H. pylori causes failure of treatment. Furazolidone, amoxicillin and tetracycline are good candidates for rescue therapy since resistance to these three antimicrobials was rare. It is necessary to assess the efficacy and safety of these four bismuth-containing quadruple regimens with above antibiotics as empirical rescue therapies for H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori -positive patients with functional dyspepsia and scarred peptic ulcers who had previously failed one or more eradication regimens containing clarithromycin, metronidazole and/or amoxicillin.

Exclusion Criteria:

* less than 18 years old, never receiving eradication treatment before, with previous gastric surgery, pregnancy, lactation, major systemic diseases, administration of antibiotics, bismuth, antisecretory drugs in the preceding 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
eradication rate of H. pylori | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liang X, Xu X, Zheng Q, Zhang W, Sun Q, Liu W, Xiao S, Lu H. Efficacy of bismuth-containing quadruple therapies for clarithromycin-, metronidazole-, and fluoroquinolone-resistant Helicobacter pylori infections in a prospective study. Clin Gastroenterol Hepatol. 2013 Jul;11(7):802-7.e1. doi: 10.1016/j.cgh.2013.01.008. Epub 2013 Jan 29. PMID 23376004